CLINICAL TRIAL: NCT03448861
Title: CHroniSense National Early Warning Score Study
Acronym: CHESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BlueWind Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP- 090
Record Dates: First submitted 2018-02-14; First posted 2018-02-28 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Clinical Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polso Wearable watch (Experimental): Polso Wearable watch for the purpose of NEWS measurement
  Interventions: Device: Polso Wearebale watch

INTERVENTIONS:
Device: Polso Wearebale watch — The objective of the Polso™ feasibility study is to demonstrate the suitability of Polso™ as a data acquisition and processing platform by comparison with the conventional British version of EWS (UK-NEWS) on aggregate and on each individual parameter score. Although in a full NEWS system, the frequency of testing is determined by the score itself, this aspect will not be evaluated, in the event that a divergence of scores would complicate clinical evaluation and correspondence of readings. In addition, good clinical practice calls for patient care to be fully motivated by the NEWS currently in use, as opposed to the experimental Polso™. Therefore, this compromise will be made, which will still permits system evaluation.

SUMMARY:
ChroniSense Medical Ltd. is developing a wearable medical multi-parametric monitoring system, Polso™. Polso™ provides a number of the parameters employed in various Early Warning Scores (EWS), such as the National Early Warning Score (NEWS), utilised widely in UK hospitals.

The EWS is a physiological track and trigger system that is generated from multi- parameter or aggregate of vital signs measurements for early recognition of clinical deterioration in acutely admitted patients. Patients who are admitted into hospital are monitored with routinely measurements of these parameters that are manually recorded on a clinical chart.

DETAILED DESCRIPTION:
ChroniSense Medical Ltd. is developing a wearable medical multi-parametric monitoring system, Polso™. Polso™ provides a number of the parameters employed in various Early Warning Scores (EWS), such as the National Early Warning Score (NEWS), utilised widely in UK hospitals.

The EWS is a physiological track and trigger system that is generated from multi- parameter or aggregate of vital signs measurements for early recognition of clinical deterioration in acutely admitted patients. Patients who are admitted into hospital are monitored with routinely measurements of these parameters that are manually recorded on a clinical chart.

The parameters of the NEWS include: 1) respiratory rate pulse rate, 2) oxygen saturations, 3) body temperature; 4) systolic blood pressure, 5) heart rate, and 6) level of consciousness. Polso™ acquires, derives, and processes a number of physiological parameters. While ECG is not currently employed in NEWS, other parameters which are used in NEWS are available in the Polso™ system. In cases where manual testing is preferred for any parameter, such as use of supplemental oxygen, the individual score can be entered into the system manually. Polso™, as a wrist-based device, could enable a degree of flexibility in patient care and management.

The goal of this study is to evaluate the suitability of Polso™ as a data acquisition and processing platform capable of providing EWS summaries, against the currently employed NEWS system at the Milton Keynes University Hospital (MKUH) Cardiology Unit. The Polso™ will be employed strictly as a data-gathering system, and will not be used to influence any clinical decisions; the standard NEWS as currently employed will fulfill all its normal clinical roles.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or female, aged 18 years or above

Exclusion Criteria:

* Unable or unwilling to give valid consent for participation in the study
* Known history of allergy to nylon
* Current diagnosis of sustained or non-sustained ventricular/atrial arrhythmia (Ventricular tachycardia, supraventricular tachycardia, atrial fibrillation, bigeminy and trigeminy)
* Weak pulse
* Patients with infectious diseases requiring isolation such as Methicillin Resistant Staphylococcus Aureus (MRSA), Clostridium difficile and Extended Spectrum Beta-Lactamases (ESBL)
* Patients with implantable defibrillators, pacemakers or neurostimulators
* Patients with Parkinson disease or essential tremor
* Patients with poor Llead I ECG signal

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
blood pressure | Through study completion, an average of 1 year
  millimeters of mercury obtained by the Polso™
pulse rate | Through study completion, an average of 1 year
  bpm obtained by the Polso™
respiratory rate | Through study completion, an average of 1 year
  number of breaths per minute obtained by the Polso™
oxygen saturation | Through study completion, an average of 1 year
  percent obtained by the Polso™
body temperature | Through study completion, an average of 1 year
  Celsius temperature scale obtained by the Polso™

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Van Velthoven MH, Adjei F, Vavoulis D, Wells G, Brindley D, Kardos A. ChroniSense National Early Warning Score Study (CHESS): a wearable wrist device to measure vital signs in hospitalised patients-protocol and study design. BMJ Open. 2019 Sep 20;9(9):e028219. doi: 10.1136/bmjopen-2018-028219. PMID 31542738